CLINICAL TRIAL: NCT05461755
Title: Treatment of Striae Distensae With Fractional Radiofrequency and Topical Tretinoin: An Intra-individual Study With Blinded Outcome Assessment
Brief Title: Treatment of Striae Distensae With Fractional Radiofrequency and Topical Tretinoin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Consultant in Dermatology, Clinical Professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDRFTT; 2021-003153-39 (EudraCT Number); H-21038853 (Other: The Regional Health Research Ethics Committee)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Striae Distensae
MeSH Terms: conditions — Striae Distensae | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, randomized and intra-individual clinical trial comparing untreated striae (controls) to striae treated with topical tretinoin and radiofrequency, respectively, and to combination therapy.
Who Masked: Outcomes Assessor
Masking Description: Primary outcome assessment is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combination therapy: Fractional radiofrequency and topical tretinoin (Experimental): 3 study treatments: at baseline, 1-month, 2-month with subsequent application of topical tretinoin. Home application of tretinoin between study visits
  Interventions: Combination Product: Fractional radiofrequency and topical Tretinoin
- Fractional radiofrequency (Active Comparator): 3 study treatments: at baseline, 1-month, 2-month
  Interventions: Device: Fractional radiofrequency
- Topical tretinoin (Active Comparator): Application at study visits and home application between study visits
  Interventions: Drug: Topical Tretinoin
- Untreated control (No Intervention): No study treatments

INTERVENTIONS:
Combination Product: Fractional radiofrequency and topical Tretinoin — Treatment of striae with fractional radiofrequency and topical tretinoin in combination
  Other Names: VenusViva MD, Retirides
  Arms: Combination therapy: Fractional radiofrequency and topical tretinoin
Drug: Topical Tretinoin — Treatment of striae with topical tretinoin alone
  Other Names: Retirides
  Arms: Topical tretinoin
Device: Fractional radiofrequency — Treatment of striae with fractional radiofrequency alone
  Other Names: VenusViva MD
  Arms: Fractional radiofrequency

SUMMARY:
The study aims to explore the potential of combination therapy with fractional radiofrequency and topical tretinoin for treatment and overall improvement of striae albae. We also aim to assess subject satisfaction, local skin responses and adverse effects/reactions in relation to the treatments, alone and in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent
2. Subject is 18 years of age or older
3. Fitzpatrick skin type I-III
4. Striae albae (grade II-IV) ≥1 year of age and ≥ 4 lesions with a length of ≥ 2 cm each
5. Women of childbearing potential are not pregnant (confirmed by a negative u-HCG prior to study treatments) and use a safe contraceptive method prior to treatments.

Exclusion Criteria:

1. Severe concurrent conditions such as cardiac disorders or poorly regulated diabetes
2. History of skin disorders such as keloids, abnormal wound healing or very fragile skin
3. History of heat-stimulated disease such as herpes simplex in the treatment area
4. History of bleeding coagulopathies or use of anti-coagulants
5. Surgery in the treatment area past 6 months or before complete healing
6. Tattoo or permanent make-up in treatment area
7. Excessively tanned skin from sun, tanning bed or tanning creams last 2 weeks
8. Dermabrasion, resurfacing, soft tissue/fat injections or chemical peeling in treatment area the past 3 months
9. Abnormal skin (e.g. rash, infection, dermatitis) at the treatment area at the time of inclusion
10. Treatment with Isotretinoin within the past 6 months
11. Use of non-steroidal anti-inflammatory drugs 1 week prior to treatment
12. Known allergies to tretinoin or lidocaine/prilocaine
13. History of cancer including pre-malignant moles
14. Impaired immune system due to immunosuppressive disease or medication
15. Electronic device implant
16. Any implantable metal piece or permanent chemical substance in treatment area
17. If female; lactating, pregnant or planning on becoming pregnant during the study
18. Non-eligibility at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Improvement in appearance of striae with GAIS | Baseline, at 4 weeks, 8 weeks and 20 weeks follow-up
  Standardized clinical photos from baseline and follow-up comparing treatments and assessed by blinded evaluator on the Global Aesthetic Improvement Scale (GAIS)

SECONDARY OUTCOMES:
Evaluation of striae with POSAS | Baseline - 20 weeks follow-up (12 weeks after last treatment)
  Standardized on-site assessment comparing treatments assessed by the subject and a blinded evaluator on the Patient-Observer Scar Assessment Scale (POSAS)
Evaluation of striae with imaging | Baseline, at 4 weeks, 8 weeks and 20 weeks follow-up
  Assessment of tissue interaction with imaging techniques
Subject satisfaction | Baseline - 20 weeks follow-up (12 weeks after last treatment)
  Likert scale for subject satisfaction
Safety: LSR and AE/AR | Baseline, at 4 weeks, 8 weeks and 20 weeks follow-up
  Collection and registration of local skin reactions and AE/AR

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD PhD DMSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Denmark